CLINICAL TRIAL: NCT03552250
Title: Prevention of Child Mental Health Problems in Southeastern Europe - Adapt, Optimize, Test and Extend Parenting for Lifelong Health
Brief Title: Prevention of Child Mental Health Problems in Southeastern Europe
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universitaet Braunschweig (Other)
Collaborators: University of Klagenfurt (Other); University of Oxford (Other); Bangor University (Other); Babes-Bolyai University (Other); Institute for Marriage, Family and Systemic Practice - ALTERNATIVA (Other); Health for Youth Association, Moldova (Other); University of Cape Town (Other); Georgia State University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Nina Heinrichs, Prof. Dr. Nina Heinrichs, Technische Universitaet Braunschweig
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H2020-779318; H2020-SC1-2017-RTD-779318 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2018-05-16; First posted 2018-06-11 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Child Mental Disorder
Keywords: Parenting Program
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parenting for Lifelong Health (Other): Parenting Programme "Parenting for Lifelong Health for Young Children" (PLH) for parents of children aged 2-9, 12 sessions
  Interventions: Behavioral: Parenting for Lifelong Health for Young Children

INTERVENTIONS:
Behavioral: Parenting for Lifelong Health for Young Children — In this study, the 12 sessions-PLH version for parents of young children (2-9 years) will be delivered. The PLH (2 - 9) programme is delivered in groups of parents and includes the following general content 1) One-on-one time, 2) Say what you see, 3) Talking about feelings, 4) Praising and rewarding our children, 5) Giving positive, specific, and realistic instructions, 6) Establishing household rules and routines, 7) Redirecting negative behavior, 8) Ignoring negative attention seeking and demanding behavior, 9) Using consequences to support compliance, 10) Using Cool-down as a consequence for aggressive behavior, 11) Avoiding and resolving conflicts, 12) Reflection celebration, and moving on.
  Other Names: PLH Programme

SUMMARY:
The aim of this study is to develop an adapted version of a low-cost parenting program (Parenting for Lifelong Health for Young Children, PLH) to the specific needs of families in three low- and middle income countries (LMICs) in southeastern Europe (Romania, FYR of Macedonia and Republic of Moldova). The investigators want systematically evaluate key barriers and facilitators at the local, national and international levels that impact prevention of child behavioral disorders.

The investigators will prepare training materials adapted to Romanian, Moldovian, Albanian, Macedonian, and Russian and train facilitators and mentor coaches in the delivery of the PLH program in each country. Also, a pre-post study will be conducted testing the feasibility of the program and the evaluation and implementation methods with 40 families at each country site. This includes examination of outcomes related to implementation fidelity, program acceptability, and preliminary program effectiveness on reducing child behavior problems and associated risk factors.

This feasibility study is part of a larger implementation project. Developed on the MOST framework (the multiphase optimization strategy), this specific study will reflect the implementation of the first phase. There are two more phases to come: the Parenting for Lifelong Health for Young Children program will be optimized within the three countries by determining which components are most efficacious and cost-effective (phase 2). The optimized PLH programs will be tested in three RCTS in the countries (phase 3).

DETAILED DESCRIPTION:
Over the past decade there have been increasing calls for the scale-up of evidence-based interventions in order to reduce the risk of violence against children in low- and middle-income countries (LMICs) (Mikton et al., 2014). In particular, parenting programs for families with young children have been shown to be effective in reducing the risk of child maltreatment and improving child wellbeing with promising evidence emerging from low- and middle-income countries (Barlow et al., 2006; Knerr et al., 2013, Chen & Chan, 2015). These group-based programs typically aim to strengthen caregiver-child relationships through positive parenting and help parents to manage child behavior problems through effective, age-appropriate, nonviolent discipline strategies.

Despite the emerging evidence of the effectiveness of parenting interventions in reducing violence against children, many local governments and service providers in LMICs face multiple challenges implementing evidence-based parenting programs in resource poor contexts (Mikton, 2012). Parenting programs are often too expensive to deliver effectively at scale in low-resource settings due to their complexity, intensity, and length (Knerr et al., 2013). Parenting programs developed and evaluated in other contexts also may not fit the local service delivery context and may require adaptation to be relevant to the local culture of families. Additional program content may also be necessary to address acute economic deprivation, high community violence, and parental distress. The process of delivery may also need to be simplified to improve participant engagement and the quality of delivery.

As a result, it is essential that programs implemented in LMICs are

1. effective at reducing violence against children,
2. integrated within the existing service delivery system,
3. feasible and culturally acceptable to service providers and families, and
4. scalable in terms of their affordability, replicability, and sustainability while reaching a maximum number of beneficiaries.

However, there are currently very few parenting programs that meet these criteria in LMICs (such as Romania, FYR of Macedonia and Republic of Moldova), where the need is the greatest.

The present study utilizes the Multiphase Optimization Strategy (MOST) as a framework for increasing the reach and enhancing the implementation of a parenting intervention for families with 2-9 years old children (Parenting for Lifelong Health for Young Children, PLH 2-9) in three southeastern European countries with restricted resources. The MOST framework is implemented over 3 distinct phases: 1) Preparation and Adaptation, 2) Optimization, and 3) Evaluation.

The Preparation and Adaptation Phase lays the foundation for program optimisation. This may include formative research, cultural/contextual adaptation, and feasibility piloting in preparation for further testing. A key objective of the Preparation Phase is to confirm the conceptual model of RISE that informs the selection of program components to optimize. Feasibility studies are considered important steps in preparation for larger experimental studies. They allow for the assessment of intervention feasibility by examining program dosage, implementation fidelity, and participant satisfaction. Although often limited in their ability to detect significant effects due to small sample sizes, feasibility studies are also opportunities to conduct exploratory analyses of intervention effects. This is particularly important when probing for potential harmful effects prior to testing in a larger population.

The RISE Study therefore includes developing three locally adapted variants of a promising parenting program which will be focused on the needs of families from LMICs with children ages 2 to 9 years who show elevated levels of externalizing problem behavior.

This feasibility study can be located in the Preparation and Adaptation phase of MOST. It is a small-scale feasibility pilot to test the feasibility of the 12-session PLH 2-9 and the evaluation and implementation methods (including preliminary outcomes of program effects). It is planned to create a locally-developed, evidence-based parenting intervention for 40 families per country. The following activities are linked to this study:

* Interviews with officials, experts and practitioners: interviews with 12-20 officials, experts and practitioners in order to gather information relating to their perceptions of the design and adaptation of a parenting intervention in;
* Gathering input from Parenting Experts Working Group in each country: meetings with a 6-member Parenting Experts Working Group, in order to incorporate these findings and their own expert opinions into the adaptation of PLH 2-9 content, process, and structure;
* Pre-Post Feasibility Study: a small-scale, pre-post evaluation to test the feasibility of the program with 40 families with children aged 2-9 years with elevated levels of child behavior problems (assessed with the Eyberg Child Behaviour Inventory, ECBI, a parent report of child externalizing problem behaviors) in each country site to examine outcomes related to implementation fidelity, program acceptability, and preliminary program effectiveness on reducing child behavior problems and associated risk factors. Moreover, the feasibility of the assessment procedures and the measures (not yet available in these regions/languages) will be tested. This means that based on the psychometric results of the feasibility study, measures may or may not be suitable for evaluation all of the listed outcomes.
* Preparation of the training materials adapted in Romanian, Moldovian, Albanian, Macedonian, and Russian, taking into account adaptation needs identified in the first three activities;
* Training of facilitators and mentor coaches in the delivery of the PLH 2-9 program in each country.

Based on the feasibility study (Adaptation and Preparation phase), the other two phases of the MOST framework will be tested in future research (studies will be registered separately):

* Phase 2: Optimization study using a factorial design testing 4 components of the parenting intervention
* Phase 3: The evaluation phase will involve testing of the optimized design (identified in phase 2) in a multisite randomised controlled trial.

A secondary objective of this project is to carefully assess barriers to implementation, integration with existing service delivery systems, and scale-ups from the outset to facilitate sustainability and real world applicability at the end of the project. When introducing such an innovative intervention in resource-limited settings, it is important to focus on the implementation processes that increase reach, efficacy, adoption, and sustainability of culturally-adapted and optimized versions of the program in addition to evaluating program effectiveness. The theoretical model for the implementation framework in the RISE project is RE-AIM (Reach, Efficacy, Adoption, Implementation, Maintenance, Glasgow et al., 2011). As a result, investigators will examine the adoption (defined as the proportion of settings willing to initiate the intervention), reach (the proportion of eligible individuals that participate in the intervention) and implementation (the fidelity, adherence, dosage assessed with multiple measures) as well as on effectiveness and sustainability of the RISE project at the organizational and participants' level. In addition, it will be examined how implementation factors influence program effectiveness, and how potential population characteristics might affect outcomes (e.g., moderators such as child age, gender, ethnicity, poverty, level of child behaviour problems, and other adversities).

ELIGIBILITY:
Inclusion Criteria:

* for caregivers/parents:

  1. age 18 or older;
  2. primary caregiver responsible for the care of a child between the ages of two and nine;
  3. Report elevated levels of child behavior problems for the child he/she chooses to be part of the study (based on the Eyberg Child Behavior Inventory);
  4. Have lived in the same household as this child at least four nights a week in the previous month and will continue to do so;
  5. agreement to participate in the PLH 2-9 program;
  6. Provision of Informed consent to participate in the full stud

Exclusion Criteria:

* for caregivers/parents: any adult 1) exhibiting severe mental health problems or acute mental disabilities; 2) that has been referred to child protection services due to child abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-12-02 (Actual)

PRIMARY OUTCOMES:
Change in levels of externalizing problem behavior in children: Child Behavior Checklist (CBCL) 11/2-5 and 6-18, parent-report, Externalizing Scale | Pre-Post (approximately 16 - 20 weeks after pre-assessment)
  The primary outcome child behavior problems is assessd with two methods: 1) parent-report: Child Behavior Checklist (CBCL). The CBCL is part of the Achenbach System of Empirically Based Assessment (ASEBA) and is available for different age ranges. For the present study, the parent-report versions for children aged 1½ - 5 and 6-18 are employed. It is the most widely used instrument for assessing child behavioral and emotional symptoms. The externalizing subscale raw score ranges from 0 to 70 (CBCL 6-18 version) and 0 to 48 (CBCL ½ - 5 version) and can be converted into standardized scores (e.g., T scores, with Mean = 50, SD = 10) with higher scores indicating more problems.
Change in Prevalence of Oppositional Defiant Disorder (ODD) and Conduct Disorder (CD)) in children: The Mini International Neuropsychiatric Interview for Children and Adolescents - Parent Version; MINI-KID-P Clinician-rated | Pre-Post (approximately 16 - 20 weeks after pre-assessment)
  The primary outcome child behavior problems is assessed with two methods: 2) structured interview, clinician-rated: The Mini International Neuropsychiatric Interview for Children and Adolescents - Parent Version; (MINI-KID-P) evaluates the presence of current psychiatric disorders (based on ICD-10 and DSM-5). It will be assessed whether or not the criteria for a) conduct disorder (F91.1, F91.2, F91.9) or b) Oppositional Defiant disorder (F91.3) are met (yes/no). The results of the two disorders will be combined to one binary total score with 0 (no externalizing disorder) and 1 (current externalizing disorder (ODD or CD)). As the sample size is small in this study phase, there is no real change in prevalence expected. However, the feasibility of the interview will be tested for later study phases with larger sample sizes.

SECONDARY OUTCOMES:
Change in levels of internalizing problem behavior in children: Child Behavior Checklist (CBCL) 11/2-5 and 6-18 parent-report, Internalizing Scale | Pre-Post (approximately 16 - 20 weeks after pre-assessment)
  Child Behavior Checklist (CBCL). The CBCL is part of the Achenbach System of Empirically Based Assessment (ASEBA) and is available for different age ranges. For the present study, the parent-report versions for children aged 1½ - 5 and 6-18 are employed. It is the most widely used instrument for assessing child behavioral and emotional symptoms. The internalizing subscale raw score ranges from 0 to 64 (CBCL/ 6 - 18 version) and 0 to 62 (CBCL/1 ½ - 5 version) and can be converted into standardized scores (e.g., T scores Mean = 50, SD = 10) with higher scores indicating more emotional problems.
Change in Prevalence of Anxiety Disorders in children: Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID-P) / Structured Clinical Diagnostic Interview for Parents, Clinician-rated | Pre-Post (approximately 16 - 20 weeks after pre-assessment)
  The Mini International Neuropsychiatric Interview for Children and Adolescents - Parent Version; (MINI-KID-P) is a structured interview to evaluate the presence of current psychiatric disorders in children (based on ICD-10 and DSM-5). It will be assessed whether or not the criteria for Separation Anxiety Disorder (F93.0), Social Anxiety Disorder (F40.1, F93.2), Specific Phobia (F40.2, F93.1), Generalized Anxiety (F41.1, F93.80) and Obsessive-Compulsive Disorder (F42.2) are currently met (yes/no). The results will be combined to one binary total score 0 (no anxiety disorder) and 1 (current anxiety disorder (criteria for at least one of the anxiety disorders met). As the sample size is small in this study phase, there is no real change in prevalence expected. However, the feasibility of the interview will be tested for later study phases with larger sample sizes.
Change in levels of psychological distress in parents: Depression, Anxiety, and Stress Scales - short version/ self-report | Pre-Post (approximately 16 - 20 weeks after pre-assessment)
  Depression, Anxiety, Stress Scales (DASS) will assess parent-report of parental depression, a 21-item scale used as a screening tool to measure depression, anxiety, and stress in adults. Caregivers report on the frequency of symptoms in the previous week using a Likert scale (0 = Never, 1 = Sometimes, 2 = Often, 3 = Always; e.g., "I felt that I had nothing to look forward to"). Total DASS scores range from 0 to 63 with subscales from 0 to 21. Recommended cut-offs indicating severity of depression are 5-6 for mild, 7-10 for moderate, 11-13 for severe, and 14 and up for extremely severe. Cut-offs for anxiety are 4-5 for mild, 6-7 for moderate, 8-9 for severe, and 10 and up for extremely severe. Cut-offs for stress are 8-9 for mild, 10-12 for moderate, 13-16 for severe, and 17 and up for extremely severe. The DASS is a widely used measure across parenting studies including those of PLH 2-9 and will allow comparison to existing results of intervention studies in non-LMICs.
Change in levels of parental well-being: WHO-5 Well-Being Scale/ self-report | Pre-Post (approximately 16 - 20 weeks after pre-assessment)
  The WHO-5 Well-Being Scale (WHO-5) will measure parental psychological well-being. This 5-item scale was derived using psychometric analyses from the longer 28-item WHO Well-Being Scale. The validation study of the WHO-5 showed 93% sensitivity and 64% specificity when compared with the General Health Questionnaire and the Patient Health Questionnaire. Parents indicate the frequency that they experienced well-being in the past month (e.g., "My daily life has been filled with things that interest me") based on a 6-point Likert scale from 0 to 5 ("At no time" to "All of the time"). Items are added up with scores ranging from 0 to 25. The Index was developed in Denmark, is very short and is available in a variety of languages, including Romanian. This scale has also been used in PLH trials in other countries and will allow comparison of results to those studies.
Change in levels of parental stress: Parenting Stress Index - Short Form (PSI-SF) / self-report | Pre-Post (approximately 16 - 20 weeks after pre-assessment)
  Parenting Stress Index-Short version (PSI-SF). The PSI-SF is a brief version (36 items) of the Parenting Stress Index. The PSI has been used extensively in parenting intervention studies and studies investigating mental health in children and their parents. It has three subscales (parental distress, parent-child dysfunctional interaction, and difficult child), and items are scored on a 5-point scale (from strongly agree to strongly disagree). Investigators will not use the Difficult Child scale due to the large overlap with the screening instrument (ECBI) and the Child Behavior Checklist; thus, the number of items used will be 24 in this study. This scale has been used in PLH trials in other countries and will allow comparison of results to those studies.
Change in incidence and frequency of child maltreatment: ISPCAN-Child Abuse Screening Tool -Intervention / self-report | Pre-Post (approximately 16 - 20 weeks after pre-assessment)
  Child maltreatment will be measured using parent report of the ISPCAN Child Abuse Screening Tool-Intervention scale (19 items, ICAST-I), an adaptation of the multi-national and consensus-based ICAST-P. The response code for the ICAST-I was adapted to a scale from 0 to more than 8 times to assess the frequency of a certain behaviour in the past month. This study will use the subscales for physical abuse, emotional abuse and neglect. The incidence of child maltreatment will be assessed by creating dichotomous variables for physical abuse, verbal abuse, and neglect, as well as an overall indication of previous child abuse (0 = no abuse; 1 = previous abuse). Investigators will also assess frequency of overall abuse by summing all of the subscales as well as for each individual subscale.
Change in frequency of dysfunctional parenting: Parenting Scale (PS) / self-report | Pre-Post (approximately 16 - 20 weeks after pre-assessment)
  The Parenting Scale (PS) was designed to explicitly measure dysfunctional discipline practices in parents. Three subscales may be derived (Laxness, Overreactivity, and Verbosity). Each item is rated on a 7-point Likert Scale by a parent ranging from 1 to 7. For computation of the subscale scores as well as the total score, the responses on the items are averaged. The range for the three subscale scores and the total score is 1 to 7 with higher scores indicating more dysfunctional parenting. The total score as well as the three subscale scores will be analysed.
Change in frequency of positive parenting and effective discipline: Parenting of Young Children Scale (PARYC) / self-report | Pre-Post (approximately 16 - 20 weeks after pre-assessment)
  Parenting of Young Children Scale (PARYC). Positive parenting behaviour will be assessed using parent-report of the Parenting of Young Children Scale (PARYC, 21 items). The PARYC measures the frequency of parent behaviour over the previous month. Items are summed to create a total frequency scores parenting behaviour as well as for the subscales: positive parenting (7 items, e.g., "how often do you play with your child"), setting limits (7 items, e.g., "how often do you stick to your rules and not change your mind") and proactive parenting (7 items, e.g., "how often do you explain what you want your child to do in clear and simple ways"). This scale has been used in PLH trials in other countries and will allow comparison of results to those studies.

OTHER OUTCOMES:
Change in levels of Intimate Partner Violence: Adapted Revised Conflict Tactics Scale-Short Form | Pre-Post (approximately 16 - 20 weeks after pre-assessment)
  Intimate partner violence will be assessed with a screening instrument, which is an adaption of the revised Conflict Tactics Scale (CTS2S). The CTS2S assesses adult self-report of exposure to intimate partner physical and psychological aggression. Assessments measure the frequency of negotiation, physical assault, psychological aggression, and physical injury. Answers are coded on a 5-point Likert scale of 0 to 4 (0 = never happened; 4 = more than 3 times in the past month), with an additional response for incidences that happened but not in the past month. This measure indicates an overall indication of IPV on a level of severity (sum of items) and prevalence (dichotomous variable indicating experience of conflict or not) as well as for each subscale.
Change in levels of family functioning, Family assessment device Short form | Pre-Post (approximately 16 - 20 weeks after pre-assessment)
  Family Assessment Device Short Form. The 12 item short form of the Family Assessment Device (FAD, General functioning) will be used to assess family functioning. The FAD is one of the most widely used instruments to assess overall family functioning. For computation of the total score, the responses on each item (ranging from 1 to 4) are averaged. Thus, the total score ranges from 1 to 4 with higher scores indicating greater family pathology.
Change in levels of parental relationship quality: Kansas Marital Satisfaction Scale | Pre-Post (approximately 16 - 20 weeks after pre-assessment)
  Kansas Marital Satisfaction Scale. This 3 item measure assesses relationship satisfaction among intimate partners. This scale has been widely used and correlates highly with other measures of relationship satisfaction (e.g., Dyadic Adjustment Scale, Quality of Marriage Index). Items are rated on a scale from 1 (extremely dissatisfied) to 7 (extremely satisfied). High internal consistency, discriminant validity, and concurrent validity have been demonstrated in other studies.
Change in levels of social community support, MOS Social Support Survey - Emotional Support Subscale, self-report | Pre-Post (approximately 16 - 20 weeks after pre-assessment)
  MOS-Social Support Survey. Perceived social support will be measured using the emotional support subscale of the Medical Outcome Study Social Support Survey (MOS-SSS, 8-items). In validation studies this scale has shown excellent internal consistency (α = 0.91 to 0.97) and test-retest reliability (α = 0.72 to 0.78). Parents report on the frequency of how often they receive emotional support (e.g., "someone you can count on to listen to when you need to talk") on a Likert-like scale of 1 to 5 (1 = none of the time; 5 = all of the time). Total scores are calculated by averaging the scores for each item and then transformed into a 0 to 100 scale. The scale was found to be distinct from related health measures, which is important for the present study.
RE-AIM Reach: Recruitment rate | Post (after 12 sessions; approximately 10-12 weeks after pre-assessment)
  Number of families who were eligible for inclusion and provided consent to participate in the program divided by the number of target population who were exposed to recruitment activities
RE-AIM Reach: Enrollment rate | Post (after 12 sessions; approximately 10-12 weeks after pre-assessment)
  Number of families who attend at least one session of the program divided by the number of families recruited into the program
RE-AIM Reach: Participation rate | Post (after 12 sessions; approximately 10-12 weeks after pre-assessment)
  Mean attendance rate for program sessions based on those families who enrolled in the program (i.e., parents who attended at least one session). Percentage of families who enrolled in the program who attended 50% (e.g., 6 sessions) and 75% (e.g., 9 sessions) or more.
RE-AIM Implementation Dosage in hours | Post (after 12 sessions; approximately 10-12 weeks after pre-assessment)
  Average number of hours delivered by facilitators (time for pre-program consultation plus session plus phone consultations per participant, facilitator report verified by implementation monitors)
RE-AIM Implementation Dosage (points of contact) | Post (after 12 sessions; approximately 10-12 weeks after pre-assessment)
  Total number of points of contact by facilitators
RE-AIM Implementation Fidelity (percentage of session activities delivered per session) | Post (after 12 sessions; approximately 10-12 weeks after pre-assessment)
  Percentage of number of session activities delivered by facilitators (by facilitator group, implementing agency, and participating country site; facilitator fidelity check-list reports verified by implementation monitors and random video recordings of session delivery)
RE-AIM Implementation Fidelity (mean percent of activities delivered per session) | Post (after 12 sessions; approximately 10-12 weeks after pre-assessment)
  Average number of activities delivered divided by total number of activities per session (by facilitator group, implementing agency, and participating country site; facilitator reports verified by implementation monitors and random video recordings of session delivery)
RE-AIM Implementation Quality | Post (after 12 sessions; approximately 10-12 weeks after pre-assessment)
  The implementation quality is assessed using the PLH-Facilitator Assessment Tool (PLH-FAT): Seven standard behaviour categories are grouped into two scales based on the core activities and process skills. Assessment of core activities includes quality of delivery during home activity review, illustrated story discussions, and practicing skills with scores from 0 (inadequate) to 3 (exceeds expectations). Assessment of process skills includes modelling skills, collaborative facilitation approach, encouragement of participation, and leadership skills (scoring from 0 = inadequate to 3 = outstanding). The total scores oft both subscales range from 0 to 72 with higher scores indicating higher facilitator competency. The total percent score for both subscales will be calculated (total score / total possible score) x 100%. A higher percent score indicates higher implementation quality.
Participants observed change in parenting practices and child behaviour at home during program | Post (approximately 16 - 24 weeks after pre-assessment)
  Qualitative in-depth interviews with intervention participants and focus groups with the facilitators in order to explore program acceptability. Participants will be purposively selected based on those with high attendance (>75%), those with low attendance (<25%), those who dropout, and those who do not enroll.
Acceptability and appropriateness of program materials, delivery, and key program components | Post (approximately 16 - 24 weeks after pre-assessment)
  Qualitative in-depth interviews with intervention participants and focus groups with the facilitators. Participants will be purposively selected session based on those with high attendance (>75%), those with low attendance (<25%), those who dropout, and those who do not enroll.
Existing barriers to participation during sessions and engagement in home practice and other activities | Post (approximately 16 - 24 weeks after pre-assessment)
  Qualitative in-depth interviews with intervention participants and focus groups with the facilitators in order to explore program acceptability. Participants will be purposively selected from the intervention group with the inclusion criteria of attending at least one intervention session. Selection will be based on those with high attendance, those with low attendance, those who dropout, and those who do not enroll.
Challenges in implementing the program | Post (approximately 16 - 24 weeks after pre-assessment)
  Qualitative focus group discussions with the facilitators exploring challenges in implementing the program on a process (e.g., using a collaborative approach and/or explaining concepts such as child led play) and logistical level (e.g., recruitment, session length, location, meals).

CONTACTS AND LOCATIONS:
Overall Officials: Heather Foran, Prof., Principal Investigator — Adria-Adria-University Klagenfurt; Jamie Lachman, Dr., Principal Investigator — University of Oxford; Frances Gardner, Prof., Principal Investigator — University of Oxford; Judy Hutchings, Prof., Principal Investigator — Bangor University; Adriana Baban, Prof., Principal Investigator — Babes Boylai University; Marija Raleva, Prof., Principal Investigator — Institute for Marriage, Family and Systemic Practice - ALTERNATIVA; Galina Lesco, Dr., Principal Investigator — Health for Youth Association, Moldova; Catherine Ward, Prof., Principal Investigator — University of Cape Town; Xiangming Fang, Prof., Principal Investigator — Georgia State University
Locations (3):
- Health For Youth Association, Chisinau, Moldova
- Institute for Marriage, Family and Systemic Practice - ALTERNATIVA, Skopje, North Macedonia
- Babes Boylai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Yes
Details will be provided in a Data Management Plan, a deliverable to the European Commission due on June 30th 2018

REFERENCES:
- [Derived] Frantz I, Foran HM, Lachman JM, Gardner F, McMahon RJ, Ogden T, Hutchings J, Costin MR, Kunovski I, Raleva M, Mueller J, Heinrichs N. Adverse event assessment in a parenting programme: experiences from a multisite randomised controlled trial. Trials. 2024 Aug 17;25(1):547. doi: 10.1186/s13063-024-08357-6. PMID 39154169
- [Derived] Frantz I, Foran HM, Lachman JM, Jansen E, Hutchings J, Baban A, Fang X, Gardner F, Lesco G, Raleva M, Ward CL, Williams ME, Heinrichs N. Prevention of child mental health problems in Southeastern Europe: a multicentre sequential study to adapt, optimise and test the parenting programme 'Parenting for Lifelong Health for Young Children', protocol for stage 1, the feasibility study. BMJ Open. 2019 Jan 25;9(1):e026684. doi: 10.1136/bmjopen-2018-026684. PMID 30782760
- See also: Project website — http://www.rise-plh.eu/index.html